CLINICAL TRIAL: NCT01167153
Title: A 12 Weeks, Multi-center, Open Label, Randomized, Active Drug Parallel Control Trial to Compare the Effectiveness of Valsartan/Amlodipine and Nifedipine in Treating Chinese Hypertensive Patients Not Respond to Mono Antihypertensive Treatment
Brief Title: Effectiveness of Valsartan/Amlodipine (EXforge®) and Nifedipine treAtment coMparison in Treating Chinese Hypertensive Patients
Acronym: EXAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489ACN02
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Hypertension
Keywords: Hypertension; Valsartan Amlodipine single pill combination; BP control; ABPM; Hypertensive patients not adequately controlled by mono antihypertensive drugs
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valsartan/amlodipine (Experimental): Valsartan/amlodipine 80/5 mg, one tablet once daily at 8:00 a.m. everyday for 12 weeks.
  Interventions: Drug: Valsartan/Amlodipine
- Nifedipine (Active Comparator): Nifedipine GITS (Gastro-Intestinal Therapeutic System ) 30 mg, one tablet once daily at 8:00 a.m. everyday for 12 weeks.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Valsartan/Amlodipine — Valsartan/Amlodipine 80/5mg single pill combination (SPC)
  Other Names: Exforge®
  Arms: Valsartan/amlodipine
Drug: Nifedipine — Nifedipine GITS (Gastro-Intestinal Therapeutic System ) 30 mg
  Other Names: Adalat
  Arms: Nifedipine

SUMMARY:
The purpose of this study was to compare the efficacy and safety of Valsartan/Amlodipine (EXforge®) with nifedipine, as well as vascular function index.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult outpatients had uncontrolled hypertension at both screening and randomization despite current antihypertensive monotherapy (initial dose of Angiotensin Receptor Blockers (ARB), Angiotensin Converting Enzyme Inhibitors (ACEI), Calcium Channel Blockers (CCB), diuretics or β receptor blocker)

Exclusion Criteria:

* Systolic BP (SBP) level ≥160 mm Hg (≥160 mm Hg in diabetics) or a diastolic BP (DBP) level ≥110 mm Hg (≥100 mm Hg in diabetics) at any time between screening and randomization.
* Patients with type 1 diabetes or poorly controlled type 2 diabetes (glycosylated hemoglobin >8.0%)
* Patients had evidence of hepatic disease or renal impairment
* Other exclusion criteria included evidence of secondary hypertension or history of cardio-vascular disease.
* Women who were pregnant, nursing, or of childbearing potential and not using acceptable contraception.

Other protocol-defined inclusion/exclusion criteria applied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Beijing, China

REFERENCES:
- [Derived] Xu SK, Zeng WF, Li Y, Chen LL, Xie JH, Wang JG. Effects of the valsartan/amlodipine combination and nifedipine gastrointestinal therapeutic system monotherapy on brachial pulse pressure and radial augmentation index in hypertensive patients. Blood Press Monit. 2021 Aug 1;26(4):251-256. doi: 10.1097/MBP.0000000000000527. PMID 33734121
- [Derived] Wang JG, Zeng WF, He YS, Chen LL, Wei M, Li ZP, Zhang BW, Li Y; EXAM Investigators. Valsartan/amlodipine compared to nifedipine GITS in patients with hypertension inadequately controlled by monotherapy. Adv Ther. 2013 Aug;30(8):771-83. doi: 10.1007/s12325-013-0048-x. Epub 2013 Aug 21. PMID 23963546

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valsartan/Amlodipine | Nifedipine
Started | 282 | 282
Intention to Treat (ITT) | 272 | 268
Completed | 264 | 249
Not Completed | 18 | 33
Not completed — Non-effective therapy | 1 | 4
Not completed — AE including clinical laboratory AE | 2 | 8
Not completed — Hypotension | 1 | 0
Not completed — Lost to Follow-up | 7 | 9
Not completed — Non-compliance to concomitant medication | 0 | 2
Not completed — Investigator initiation withdrawal,Other | 1 | 1
Not completed — Withdrawal consent | 1 | 1
Not completed — Subject initiation withdrawal, Other | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan/Amlodipine | Nifedipine | Total
Number analyzed (Participants) | 272 | 268 | 540
Age Continuous [Mean (Standard Deviation); unit: years] — demographic measures were based on intent to treat (ITT) population. One patient was missing from Nifedipine arm for Age, continuous measurement.
  years | 53.8 (8.59) | 53.1 (8.72) | 53.5 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 135 | 270
  Male | 137 | 133 | 270

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) at the Study End Point (12 Weeks)
Description: The sitting blood pressure was trough value (23-26 hours after drug administration) measured by sphygmomanometer. Blood pressure was measured on both arms and the arm with higher mean sitting diastolic blood pressure (MSDBP) was used at visit 1 and following visits. Measurement of blood pressure was carried out 3 times at each visit on the selected arm. The results and mean value of three sitting blood pressures were recorded for analysis.
Time Frame: Baseline, 12 weeks
Population: ITT (intention to treatment) population: all randomised subjects who had baseline assessment and at least one assessment record of MSSBP after baseline.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/Amlodipine | Nifedipine
Number analyzed (Participants) | 267 | 265
mm Hg | -16.8 (11.69) | -10.6 (12.02)

2. Primary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP) at the Study End Point (12 Weeks)
Description: The sitting blood pressure was trough value (23-26 hours after drug administration) measured by sphygmomanometer. Blood pressure was measured on both arms and the arm with higher msDBP was used at visit 1 and following visits. Measurement of blood pressure was carried out 3 times at each visit on the selected arm. The results and mean value of three sitting blood pressures were recorded for analysis.
Time Frame: Baseline, 12 weeks
Population: ITT (intention to treatment) population: all randomised subjects who had baseline assessment and at least one assessment record of MSDBP after baseline.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/Amlodipine | Nifedipine
Number analyzed (Participants) | 267 | 265
mm Hg | -8.5 (8.52) | -4.8 (8.89)

3. Secondary Outcome: Percentage of Patients With Effective Systolic Blood Pressure (SBP) Control Rate and Effective Diastolic Blood Pressure (DBP) Control Rate at the Study End Point (12 Weeks)
Description: Effective SBP control rate was defined as proportion of subjects in whom MSSBP < 140 mmHg or MSSBP reduction ≥ 20 mmHg from baseline.
  Effective DBP control rate was defined as proportion of subjects in whom MSDBP < 90 mmHg or MSDBP reduction ≥10 mmHg from baseline.
Time Frame: Baseline, 12 weeks
Population: ITT (intention to treatment) population: all randomised subjects who had baseline assessment and at least one assessment record of effective BP control after baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Valsartan/Amlodipine | Nifedipine
Number analyzed (Participants) | 267 | 265
Percentage of participants
  Achieving Effective SBP Control | 82.40 | 63.40
  Achieving Effective DBP Control | 92.88 | 76.98

4. Secondary Outcome: Percentage of Patients in Whom Blood Pressure Target Was Achieved at the Study End Point at 12 Weeks
Description: Blood Pressure (BP) target was defined as mean sitting BP<140/90 mm Hg in non-diabetic patients and<130/80 mm Hg in diabetic patients at 12 weeks.
Time Frame: 12 weeks
Population: ITT (intention to treatment) population: all randomised subjects who had baseline assessment and at least one assessment record of blood pressure control after baseline
Measure: Number; unit: Percentage of participants
Arm/Group | Valsartan/Amlodipine | Nifedipine
Number analyzed (Participants) | 267 | 265
Percentage of participants | 79.03 | 57.36

5. Secondary Outcome: Change From Baseline in Orthostatic SBP and DBP at 12 Weeks
Description: The arm with higher sitting blood pressure was selected for all examinations throughout the study. Orthostatic blood pressure was measured when subject stood for 1 minute. Orthostatic blood pressures were measured at screening and each visit.
Time Frame: Baseline, 12 weeks
Population: ITT (intention to treatment) population: all randomised subjects who had baseline assessment and at least one assessment record of orthostatic SBP and DBP after baseline.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan/Amlodipine | Nifedipine
Number analyzed (Participants) | 266 | 265
mm Hg
  Orthostatic diastolic blood pressure | -7.2 (9.43) [-8.2172 to -6.2177] | -3.3 (9.58) [-4.2475 to -2.2442]
  Orthostatic systolic blood pressure | -13.3 (13.86) [-14.3985 to -11.4312] | -8.6 (13.98) [-10.4851 to -7.5122]

6. Secondary Outcome: Change From Baseline in Sitting Pulse at 12 Weeks
Description: Sitting pulse was measured by sphygmomanometer after subject sat for 5 minutes at clinic during each visit.
Time Frame: Baseline, 12 weeks
Population: ITT (intention to treatment) population: all randomised subjects who had baseline assessment and at least one assessment record of sitting pulse rate after baseline.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Valsartan/Amlodipine | Nifedipine
Number analyzed (Participants) | 267 | 264
beats/min | -1.1 (8.49) | 0.0 (8.22)

7. Secondary Outcome: Change From Baseline in Orthostatic Pulse at 12 Weeks
Description: Orthostatic pulse was measured by sphygmomanometer when subject stood for 1 minute at clinic during each visit.
Time Frame: Baseline, 12 weeks
Population: ITT (intention to treatment) population: all randomised subjects who had baseline assessment and at least one assessment record of orthostatic pulse rate after baseline.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Valsartan/Amlodipine | Nifedipine
Number analyzed (Participants) | 266 | 264
beats/min | -0.6 (8.93) | 0.4 (8.48)

ADVERSE EVENTS:
Description: Safety analysis population: all randomised subjects who administrated at least one dose of investigational drug.
Arm/Group | Valsartan/Amlodipine | Nifedipine
Serious Adverse Events (participants affected / at risk) | 0/282 | 1/282
Other Adverse Events (participants affected / at risk) | 14/282 | 32/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan/Amlodipine (N=282) | Nifedipine (N=282)
Unstable Blood Pressure (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan/Amlodipine (N=282) | Nifedipine (N=282)
Dizzy (Nervous system disorders) | 11 | 15
Headache (Nervous system disorders) | 6 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.